CLINICAL TRIAL: NCT04068194
Title: A Phase I/II Study of M3814 and Avelumab in Combination With Hypofractionated Radiation in Patients With Advanced/Metastatic Solid Tumors and Hepatobiliary Malignancies
Brief Title: Testing the Combination of New Anti-cancer Drug Peposertib With Avelumab and Radiation Therapy for Advanced/Metastatic Solid Tumors and Hepatobiliary Malignancies
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Scheduled Interim Monitoring
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-05373; NCI-2019-05373 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 052002; 10276 (Other: Dana-Farber - Harvard Cancer Center LAO); 10276 (Other: CTEP); UM1CA186644 (NIH); UM1CA186716 (NIH)
Record Dates: First submitted 2019-08-15; First posted 2019-08-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Malignant Solid Neoplasm; Locally Advanced Unresectable Cholangiocarcinoma; Locally Advanced Unresectable Gallbladder Carcinoma; Locally Advanced Unresectable Malignant Solid Neoplasm; Metastatic Cholangiocarcinoma; Metastatic Gallbladder Carcinoma; Metastatic Malignant Solid Neoplasm; Stage III Gallbladder Cancer AJCC v8; Stage IV Gallbladder Cancer AJCC v8; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms; Neoplasm Metastasis | interventions — avelumab; Biopsy; Specimen Handling; Radiation Dose Hypofractionation; Radiation; peposertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (hypofractionated RT, avelumab) (Active Comparator): Patients undergo 8 fractions of hypofractionated RT QD on days -17 to -7. Patients also receive avelumab IV over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy, CT, and collection of blood on the trial.
  Interventions: Drug: Avelumab; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: Hypofractionated Radiation Therapy
- Arm B (hypofractionated RT, peposertib, avelumab) (Experimental): Patients undergo 8 fractions of hypofractionated RT QD on days -17 to -7. Patients also receive peposertib PO BID on days 1-28, and avelumab IV over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy, CT, and collection of blood on the trial.
  Interventions: Drug: Avelumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: Hypofractionated Radiation Therapy; Drug: Peposertib
- Phase I (hypofractionated RT, peposertib, avelumab) (Experimental): Patients with advanced/metastatic malignant solid tumors undergo 8 fractions of hypofractionated RT QD on days -17 to -7. Patients also receive peposertib PO BID on days 1-28, and avelumab IV over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, biopsy, and collection of blood samples during screening and on study.
  Interventions: Drug: Avelumab; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: Hypofractionated Radiation Therapy; Drug: Peposertib

INTERVENTIONS:
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB 0010718C; MSB-0010718C; MSB0010718C
Procedure: Biopsy Procedure — Undergo biopsy of tumor
  Other Names: Biopsy; BIOPSY_TYPE; Bx
  Arms: Arm A (hypofractionated RT, avelumab); Phase I (hypofractionated RT, peposertib, avelumab)
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated RT
  Other Names: Hypofractionated; Hypofractionated Radiotherapy; hypofractionation; Radiation, Hypofractionated
Drug: Peposertib — Given PO
  Other Names: 3-Pyridazinemethanol, alpha-(2-Chloro-4-fluoro-5-(7-(4-morpholinyl)-4-quinazolinyl)phenyl)-6-methoxy-, (alphaS)-; M 3814; M-3814; M3814; MSC 2490484A; MSC-2490484A; MSC2490484A; Nedisertib
  Arms: Arm B (hypofractionated RT, peposertib, avelumab); Phase I (hypofractionated RT, peposertib, avelumab)

SUMMARY:
This phase I/II trial studies the best dose and side effects of peposertib and to see how well it works with avelumab and hypofractionated radiation therapy in treating patients with solid tumors and hepatobiliary malignancies that have spread to other places in the body (advanced/metastatic). Peposertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as avelumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Giving peposertib in combination with avelumab and hypofractionated radiation therapy may work better than other standard chemotherapy, hormonal, targeted, or immunotherapy medicines available in treating patients with solid tumors and hepatobiliary malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability and recommended phase 2 dose (RP2D) of peposertib (M3814) in combination with hypofractionated radiation and avelumab in patients with advanced/metastatic solid tumors. (Phase I) II. To determine the efficacy of the combination of hypofractionated radiation, peposertib (M3814), and avelumab as compared to the combination of hypofractionated radiation and avelumab in patients with advanced/metastatic hepatobiliary tumors by objective response rate (ORR) in non-irradiated lesions within 12 weeks following initiation of study treatment. (Phase II)

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. (Phase I) II. To characterize the pharmacokinetic (PK) profile of peposertib (M3814) in combination with avelumab. (Phase I) III. To determine the efficacy and safety of the combination of hypofractionated radiation, peposertib (M3814), and avelumab as compared to hypofractionated radiation and avelumab by measurement of disease control rate (DCR), duration of response (DOR), progression free survival (PFS), PFS outside the irradiated field, and overall survival (OS) in patients with advanced/metastatic hepatobiliary tumors. (Phase II) IV. To determine if baseline deoxyribonucleic acid (DNA) repair defects inherent to some cholangiocarcinomas correlate with a more dramatic response to radiation compared to those without as measured by gamma H2AX, phosphorylated (p)NBS1 and pKAP1 immunofluorescence (IFA) with beta CATN segmentation assay. (Phase II) V. To characterize the pharmacokinetic (PK) profiles of peposertib (M3814) and avelumab. (Phase II)

EXPLORATORY OBJECTIVES:

I. To perform molecular profiling assays on malignant and normal tissues, including, but not limited to, whole exome sequencing (WES), ribonucleic acid (RNA) sequencing (RNAseq), mass cytometry (CyTOF), multiplexed ion beam imaging (MIBI), and T cell receptor sequencing in order to:

Ia. To determine if baseline tumor mutation burden and pattern, and neoantigen burden correlate with response; Ib. To determine if combination therapy results in changes in the immune landscape in both the tumor and the host that correlate with response; Ic. To determine if baseline defects in deoxyribonucleic acid (DNA) damage repair in some cholangiocarcinomas correlate with an increased response.

OUTLINE: This is a phase I, dose-escalation study of peposertib followed by a phase II study.

PHASE I:

Patients with advanced/metastatic malignant solid tumors undergo 8 fractions of hypofractionated radiation therapy (RT) every day (QD) on days -17 to -7. Patients also receive peposertib orally (PO) twice daily (BID) on days 1-28, and avelumab intravenously (IV) over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT), biopsy, and collection of blood samples during screening and on study.

PHASE II: Patients with advanced/metastatic cholangiocarcinoma/gallbladder cancer are randomized to 1 of 2 arms.

ARM A: Patients undergo 8 fractions of hypofractionated RT QD on days -17 to -7. Patients also receive avelumab IV over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, biopsy, and collection of blood samples during screening and on study.

ARM B: Patients undergo 8 fractions of hypofractionated RT QD on days -17 to -7. Patients also receive peposertib PO BID on days 1-28, and avelumab IV over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, biopsy, and collection of blood samples during screening and on study

After completion of study treatment, patients are followed up at 30 days, every 3 months for 1 year, every 6 months for year 2, then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* PHASE 1: Patients must have a histologically confirmed metastatic or locally advanced unresectable solid tumor that has progressed on or after available standard of care therapy or for which no acceptable standard of care therapy exists, or in which the patient declines standard of care therapy (each patient that declines standard of care therapy will be documented in the case report form)
* PHASE 2: Patients must have a histologically confirmed metastatic or locally advanced unresectable cholangiocarcinoma/gallbladder carcinoma that has progressed on gemcitabine, cisplatin, and durvalumab/pembrolizumab
* Age >= 18 years

  * Because no dosing or adverse event data are currently available on the use of peposertib (M3814) in combination with avelumab in patients < 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Patients with at least 1 index lesion to irradiate for whom palliative radiation treatment is indicated (including but not limited to pain and/or symptom control, prevention of disease -related complications, and preservation of organ function). Lung and liver lesions are preferred, though alternate lesions may be considered after discussion with trial principal investigator (PI). Up to 2 lesions may be considered for irradiation provided at least 1 lesion will receive the study treatment of total of 60 Gy and all prescribed irradiation will be completed within the radiation window
* Patients with at least 1 Response Evaluation Criteria in Solid Tumors (RECIST) measurable lesion (to be unirradiated) (defined as those accurately measured in at least one dimension, with the longest diameter to be recorded for non-nodal lesions and the shortest diameter for nodal lesions). Measurable is defined as at least 10 mm in longest diameter for solid tumors, at least 15 mm in shortest diameter for lymph nodes
* Patients must be willing to undergo fresh biopsies at baseline (as opposed to using archival tissue), in the event their baseline tissue was obtained > 12 months prior to study consent and/or they are randomized to the gamma H2AX, pNBS1 and pKAP1 IFA with beta CATN segmentation assay
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelet count >= 100,000/mcL
* Hemoglobin >= 9.0 g/dL
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR calculated serum creatinine clearance (glomerular filtration rate [GFR] can be used in place of creatinine or creatinine clearance) >= 60 mL/min for participants with creatinine levels > 1.5 x institutional ULN

  * Calculate serum creatinine clearance using the standard Cockcroft-Gault formula
* Serum total bilirubin =< 1.5 x ULN or direct bilirubin =< ULN for participants with total bilirubin > 1.5 x ULN

  * Patients with known Gilbert disease with serum bilirubin level =< 3 x ULN are eligible
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN or =< 5.0 x ULN for patients with hepatobiliary tumors/liver metastases
* Albumin >= 2.8 g/L
* International normalized ratio (INR) or prothrombin time (PT) or activated partial thromboplastin time (aPTT) =< 1.5 x ULN

  * This applies only to patients not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose
* Participants must have the ability to swallow and retain oral medication and not have any clinically significant gastrointestinal abnormalities that might alter absorption
* Female patients of childbearing potential must have a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The effects of peposertib (M3814) and avelumab on the developing human fetus are unknown and there is the potential for teratogenic or abortifacient effects. For this reason, women and men of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study treatment, and for 6 months after completion of peposertib (M3814) and avelumab administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with peposertib (M3814) and avelumab, breastfeeding should be discontinued if the mother is treated with peposertib (M3814) and avelumab
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a close caregiver or legally authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* PHASE I: Patients who have received prior anti-CTLA-4, anti-PD-1, anti-PD-L1 or other immune checkpoint inhibitor therapeutic antibodies or pathway-targeting agents
* PHASE II: Patients who have received prior anti-CTLA-4, anti-PD-1, anti-PD-L1 or other immune checkpoint inhibitor therapeutic antibodies or pathway-targeting agents with the following exceptions:

  * Patients who have only received previous durvalumab (anti-PD-L1) in combination with gemcitabine +/- cisplatin as part of first line therapy (TOPAZ-1 regimen) are eligible
  * Patients who have only received previous pembrolizumab (anti-PD-1) in combination with gemcitabine +/- cisplatin as part of first line therapy (KEYNOTE-966 regimen) are eligible
* Patients who have had chemotherapy, definitive radiation, biological cancer therapy, or investigational agent/device within 21 days of first planned dose of study therapy (within 14 days for palliative radiation). Previously irradiated lesions may be re-irradiated provided there is disease progression in the irradiated lesion and the prescribed radiation dosage can safely be re- administered
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Common Terminology Criteria for Adverse Events [CTCAE] grade 1) with the exception of alopecia
* Patients with untreated/uncontrolled central nervous system (CNS)/leptomeningeal disease. Patients with asymptomatic, treated CNS disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy and the following criteria are met:

  * Radiographic demonstration of clinical stability upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study done >= 4 weeks from completion of radiotherapy and >= 2 weeks from discontinuation of corticosteroids
  * No stereotactic radiation or whole-brain radiation within 28 days prior to randomization
* Patients with active autoimmune disease requiring systemic corticosteroids greater than the equivalent of prednisone 10 mg daily including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, colitis, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis, with the following exceptions:

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen are eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only who require only low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%) are eligible
* Patients receiving treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 6 weeks must discontinue these medications prior to starting peposertib (M3814) and avelumab, with the exception of:

  * Patients with active autoimmune disease managed with systemic corticosteroids less than the equivalent of prednisone 10 mg daily
  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea)
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension and adrenocortical insufficiency
* Patients who have undergone prior solid organ or bone marrow transplant with the exception of patients with prior renal transplant for whom dialysis may be employed in the event of graft rejection
* Patients with uncontrolled intercurrent illness (e.g., including but not limited to uncontrolled hypertension [HTN] [systolic blood pressure (BP) > 150, diastolic BP > 100], symptomatic congestive heart failure [CHF], unstable angina pectoris, ischemic myocardial infarction [MI] within 6 months, cardiac arrhythmia, transient ischemic attack [TIA or cerebrovascular accident (CVA)]) within 6 months
* Patients with serious active infection (e.g. requiring hospitalization and/or intravenous [IV] antibiotics) within 4 weeks prior to starting peposertib (M3814) and avelumab, or signs/symptoms of infection or receiving oral or IV antibiotics for the treatment of active systemic infection within 2 weeks prior to starting peposertib (M3814) and avelumab. Patients receiving prophylactic antibiotics are eligible
* Patients with known chronic hepatitis B virus (HBV) infection must have an undetectable viral load on suppressive therapy if indicated. Patients with known chronic hepatitis C (HCV) infection must have been treated and cured. Patients who are currently on curative treatment are eligible if they have an undetectable HCV viral load
* Patients with known human immunodeficiency virus (HIV) are allowed on study provided they have:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infection
  * A CD4 count above 250 cells/mcL
  * An undetectable HIV viral load on standard polymerase chain reaction (PCR)-based testing
* Patients with history of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (e.g., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Patients with known concurrent malignancy that is expected to require active treatment within two years, or may interfere with the interpretation of the efficacy and safety outcomes of this study in the opinion of the treating investigator. Superficial bladder cancer, nonmelanoma skin cancers, and low-grade prostate cancer not requiring cytotoxic therapy should not exclude participation in this trial. Patients with chronic lymphocytic leukemia (CLL) may be enrolled if they do not require active chemotherapy and their hematologic, renal and hepatic function meets criteria previously mentioned
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to peposertib (M3814) or avelumab
* Patients unable to discontinue medications or substances that are potent inhibitors, inducers or sensitive substrates of CYP3A4/5 or CYP2C19 prior to starting peposertib (M3814) and avelumab are ineligible. Medications or substances that are strong inhibitors of CYP3A4/5 or CYP2C19 must be discontinued at least 1 week prior to first peposertib (M3814) dose. Strong inducers of CYP3A4/5 or CYP2C19 must be stopped at least 3 weeks prior to the first dose. Drugs mainly metabolized by CYP3A with a narrow therapeutic index as judged by the investigator must stop at least 1 day prior to first peposertib (M3814) dose. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product. The primary elimination mechanism of avelumab is proteolytic degradation, thus there are no contraindicated medications with respect to avelumab
* Patients who cannot discontinue concomitant proton-pump inhibitors (PPIs) prior to starting peposertib (M3814) and avelumab. These must be discontinued >= 5 days prior to starting peposertib (M3814) and avelumab. Patients do not need to discontinue calcium carbonate. H2 blockers are allowed provided they are taken at least 2 hours after peposertib (M3814) dose
* Patients receiving sorivudine or any chemically related analogues (such as brivudine) and not able to discontinue prior to starting peposertib (M3814) and avelumab are excluded
* Pregnant and lactating women are excluded from this study because peposertib (M3814) and avelumab are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with peposertib (M3814) and avelumab, breastfeeding should be discontinued if the mother is treated with peposertib (M3814) and avelumab
* Patients who have received live vaccination within 30 days before starting peposertib (M3814) and avelumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2020-04-07 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated doses and recommended phase 2 dose of peposertib (M3814) in combination with hypofractionated radiation and avelumab (Phase 1) | Up to 28 days
  Will be determined by the occurrence of dose-limiting toxicities defined as the occurrence of one or more grade 3 adverse events that delays treatment for more than 7 days, or any grade 4-5 adverse events.
Objective response rate (Phase 2) | Within 12 weeks following initiation of study treatment
  Defined as best overall response (compete response [CR] and partial response [PR] in non-irradiated lesions as opposed to stable disease [SD] or progressive disease) within 12 weeks following initiation of study treatment by Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

SECONDARY OUTCOMES:
Pharmacokinetics of avelumab (Phase 1) | Day 7: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours; Day 21: predose, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours
  Will determine concentrations of plasma avelumab using enzyme-linked immunosorbent assay.
Pharmacokinetics of M3814 (Phase 1) | Day 21: predose
  Will determine concentrations of plasma M3814 using liquid chromatography-mass spectrometry (MS)/MS.
Disease control rate (Phase 2) | Up to 12 months
  Defined as proportion of patients achieving a CR, PR, or SD in non-irradiated by RECIST 1.1 criteria. Will be analyzed by Kaplan-Meier estimates.
Progression free survival (PFS) (Phase 2) | From randomization until disease progression or death, assessed up to 12 months
  Will be analyzed by Kaplan-Meier estimates.
PFS outside the irradiated field (Phase 2) | From randomization until disease progression outside the irradiated field or death, assessed up to 12 months
  Will be analyzed by Kaplan-Meier estimates.
Overall survival (Phase 2) | From randomization until death from any cause, assessed up to 12 months
  Will be analyzed by Kaplan-Meier estimates.
Incidence of adverse events (Phase 2) | Up to 12 months
  Defined by Common Terminology Criteria for Adverse Events version 5.0.
Pharmacokinetics of M3814 and avelumab (trough levels) (Phase 2) | M3814 and avelumab: Day 21 (Predose)
  Correlated with pharmacodynamics (e.g. toxicity). Will compare trough values between patients with and without toxicity, and/or response if warranted, with non-parametric testing.
Defects in deoxyribonucleic acid (DNA) damage repair | Up to 12 months
  Assessed by the gamma H2AX phosphorylated (p)NBS1 multiplex immunofluorescence assay (IFA). The association of baseline DNA repair defects, scored as present or absent, with the response rate to treatment will be evaluated using Fisher's exact test.
Differential response to therapy (Phase 2) | Up to 12 months
  Assessed by the gamma H2AX pNBS1 multiplex IFA. The association of baseline DNA repair defects, scored as present or absent, with the response rate to treatment will be evaluated using Fisher's exact test.

OTHER OUTCOMES:
Tumor mutation burden | Baseline
  Assessed by whole exome sequencing (WES). Correlates will be summarized using descriptive statistics. The association of tumor mutation scored as high or low, with response rates to treatment will be evaluated using Fisher's exact test.
Tumor mutation burden | Baseline
  Assessed by ribonucleic acid sequencing (RNAseq). Correlates will be summarized using descriptive statistics. The association of tumor mutation scored as high or low, with response rates to treatment will be evaluated using Fisher's exact test.
Tumor pattern | Baseline
  Assessed by WES. Correlates will be summarized using descriptive statistics. The association of tumor mutation scored as high or low, with response rates to treatment will be evaluated using Fisher's exact test.
Tumor pattern | Baseline
  Assessed by RNAseq. Correlates will be summarized using descriptive statistics. The association of tumor mutation scored as high or low, with response rates to treatment will be evaluated using Fisher's exact test.
Neoantigen burden | Up to 12 months
  Assessed by WES. Correlates will be summarized using descriptive statistics. The association of neoantigen burdens, scored as high or low, with response rates to treatment will be evaluated using Fisher's exact test.
Neoantigen burden | Up to 12 months
  Assessed by RNAseq. Correlates will be summarized using descriptive statistics. The association of neoantigen burdens, scored as high or low, with response rates to treatment will be evaluated using Fisher's exact test.
Defects in DNA damage repair | Baseline up to 12 months
  Assessed by WES. Immune-response gene expressions will be measured pre- and post-therapy, and be compared using a paired t-test, or a Wilcoxon signed rank test where appropriate.
Differential response to therapy | Baseline up to 12 months
  Assessed by WES. Immune-response gene expressions will be measured pre- and post-therapy, and be compared using a paired t-test, or a Wilcoxon signed rank test where appropriate.
Tumor infiltrating lymphocyte quantification and characterization | Up to 12 months
  Assessed by multiplexed ion beam imaging in both the tumor and the host.
Circulating T lymphocyte quantification and characterization | Up to 12 months
  Assessed by mass cytometry in both the tumor and the host.
T cell receptor (TCR) clonality | Up to 12 months
  Assessed by TCR sequencing in both the tumor and the host.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen R Spencer, Principal Investigator — Laura and Isaac Perlmutter Cancer Center at NYU
Locations (46):
- United States (46):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Bellevue Hospital Center, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm